CLINICAL TRIAL: NCT01061632
Title: Effects of High(Deadlift) Versus Low Intensity Motor Control Exercises on Patients With Peripherally Mediated Low Back Pain
Brief Title: High(Deadlift) Versus Low Intensity Motor Control Exercises on Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Luleå Tekniska Universitet (Other)
Collaborators: Umeå University (Other); Norrlandskliniken (Unknown); County Council of Norrbotten, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LTU_marklyft
Record Dates: First submitted 2010-01-20; First posted 2010-02-03 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Low Back Pain
Keywords: deadlift; motor control; exercises; pain; function; functional capacity
MeSH Terms: conditions — Low Back Pain; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: High intensity motor control exercise (deadlift) — 12 treatment sessions over a 8 week period is planned for the high intensity motor control exercise.
Procedure: Low intensity motor control exercise — 12 sessions of low intensity motor control exercises over 8 weeks

SUMMARY:
The aim of the study is to evaluate and compare the effects of high-intensity (deadlift) versus low-intensity motor control exercises on selfrated pain, function and symptoms on patients with peripherally mediated pain

ELIGIBILITY:
Inclusion Criteria:

* low back pain over 3 month
* the pain must originate locally from the lowe back and be nociceptive

Exclusion Criteria:

-

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Selfrated function, symptoms and pain-rating | 8 weeks, 6 month, 12 month

SECONDARY OUTCOMES:
Functional capacity | 8 weeks, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Öhrling, As professor, Study Director — Luleå Tekniska Universitet

REFERENCES:
- [Derived] Aasa B, Berglund L, Michaelson P, Aasa U. Individualized low-load motor control exercises and education versus a high-load lifting exercise and education to improve activity, pain intensity, and physical performance in patients with low back pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2015 Feb;45(2):77-85, B1-4. doi: 10.2519/jospt.2015.5021. PMID 25641309
- [Derived] Berglund L, Aasa B, Hellqvist J, Michaelson P, Aasa U. Which Patients With Low Back Pain Benefit From Deadlift Training? J Strength Cond Res. 2015 Jul;29(7):1803-11. doi: 10.1519/JSC.0000000000000837. PMID 25559899